CLINICAL TRIAL: NCT03052686
Title: Retrospective Study of 110 Cases of Uterine Rupture to Determine Obstetric and Neonatal Complications
Acronym: RUVO
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0914
Record Dates: First submitted 2016-09-13; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Anomaly Uterus
Keywords: Uterine rupture
MeSH Terms: conditions — Uterine Anomalies; Uterine Rupture | interventions — Parturition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Childbirth with uterine rupture: No intervention. Follow-up of women with uterine rupture at the childbirth.
  Interventions: Other: Childbirth with uterine rupture

INTERVENTIONS:
Other: Childbirth with uterine rupture — No intervention. Follow-up of women with rupture uterine at the childbirth.

SUMMARY:
This study has for objective to collect medical data from patients with uterine rupture at the childbirth.

DETAILED DESCRIPTION:
This is a retrospective study, gathering data of five maternity in the department of Val d'Oise in France, during 13 years (between 01/01/2000 an 31/12/2013).

The incidence of uterine rupture increases with increasing cesarean rates. It occurs at a rate of 0.08% across all childbirths in France, and 0.5 to 1% of the childbirths on cicatricial uterus in France.

Although the risk factors are known, it is usually unexpected. This is a serious complication for the mother (mortality <1%, severe morbidity at 15% ) and for the child (mortality for 3 to 6 % for childbirth at term, neonatal asphyxia for 6 to 15%) that can occur during pregnancy or during labor.

ELIGIBILITY:
Inclusion Criteria:

* Childbirth with uterine rupture

Exclusion Criteria:

* Childbirth in a maternity which do not participate to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with rupture uterine at the childbirth.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2000-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Identify maternal and foetal risk factors associated to an uterine rupture ; by the report of events during pregnancy, pathology, lifestyle, Concomitant pathology... | 1 day

SECONDARY OUTCOMES:
Number of maternal and foetal adverse events associated to an uterine rupture at the childbirth. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: MARKOU Georges, PH, Principal Investigator — CH Rene Dubos, Pontoise

IPD SHARING:
Plan to Share IPD: No